CLINICAL TRIAL: NCT05321706
Title: DAPARHT: DAPAgliflozin for Renal Protection in Heart Transplant Recipients
Brief Title: DAPAgliflozin for Renal Protection in Heart Transplant Recipients
Acronym: DAPARHT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Erasmus Medical Center (Other); Skane University Hospital (Other); Aarhus University Hospital (Other); Karolinska University Hospital (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lars Gullestad, Professor, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-003175-34
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Heart Transplant Failure; Kidney Failure
Keywords: Renal protection; Heart transplant; Dapagliflozin
MeSH Terms: conditions — Renal Insufficiency | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: The DAPARHT trial is a randomised, controlled, double blind, parallel group trial with an open-label extension phase. The primary endpoint is the slope of the eGFR measured from 2 weeks after randomisation and start of treatment to 12 months after start of treatment. The trial subjects immediately continue into the open-label phase. In this phase, patients assigned to dapagliflozin continue treatment for another 24 months. The primary endpoint of the open-label extension is the baseline-adjusted eGFR measured one month after the end of treatment, 37 months after randomisation.
Who Masked: Participant, Care Provider
Masking Description: One year's blinded treatment + two years' open-label extension. The primary endpoint of the blinded phase of the trial is the difference in the slope from 2 weeks to 12 months in the eGFR. The major endpoint of the open-label phase is the baseline-adjusted eGFR measured 1 months after the end of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): Participants will be randomized in a 1:1 fashion to receive 10 mg of oral dapagliflozin (tablet) once daily for one year.
  Interventions: Drug: Dapagliflozin 10 mg
- Placebo (Placebo Comparator): Participants will be randomized in a 1:1 fashion to receive a matching tablet once daily for one year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Participants will be randomized in a 1:1 fashion to receive 10 mg of oral dapagliflozin
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Placebo — Participants will be randomized in a 1:1 fashion to receive a matching placebo once daily for one year.
  Arms: Placebo

SUMMARY:
Kidney failure is common in heart transplant recipients and is a major cause of morbidity and mortality. Sodium-glucose transporter 2 (SGLT2) inhibitors were developed as antidiabetics but were subsequently shown to reduce the incidence of adverse cardiovascular outcomes and protect renal function in non-diabetics as well as diabetics. However, SGLT2 inhibitors have not been tested in clinical trials in heart transplant recipients. The DAPARHT trial is designed to assess the effect of the SGLT2 inhibitor dapagliflozin to prevent deteriorating renal function in heart transplant recipients. Secondary objectives are to assess the impact of treatment on i) weight, ii) glucose homeostasis, iii) proteinuria, iv) the number of rejections, and (v) safety and tolerability. As exploratory outcomes, the investigators will assess the effect of treatment on renal outcomes, clinical events (death, myocardial infarction, cerebral stroke, cancer, and end-stage renal disease), cardiac function, quality of life, and new-onset diabetes.

DETAILED DESCRIPTION:
Heart transplant is the treatment of choice for selected patients with end-stage heart failure. Worldwide, approximately 5000 procedures are performed annually. Whereas the first successful heart transplant led to a mere 18 days' prolongation of the recipient's life, the median survival after transplantation is now more than 11 years. Important surgical advances, as well as optimal medical therapy, are responsible for this improvement, but reducing morbidity and mortality further is a significant challenge. Beyond the first year, outcomes have not improved over the last decades. An important reason for this is the considerable burden of long-term side effects induced by immunosuppressive therapy. Chronic renal failure occurs in approximately 11 % of heart transplant recipients during the first five years after transplant and is associated with a large increase in mortality. A major cause of renal injury is a calcineurin inhibitor (CNI)-related nephrotoxicity. Calcineurin inhibitors revolutionized transplant medicine when introduced in the early 1980'ies and remain the mainstay of immunosuppressive therapy after a heart transplant. However, the therapy is an important contributor to post-transplant nephropathy. Furthermore, CNIs seem to contribute to metabolic disturbances including diabetes mellitus, hypertension, and oxidative stress after a heart transplant.

The deterioration of renal function after a heart transplant appears to be linear. In a Swedish material, the average yearly drop in the estimated glomerular filtration rate (eGFR) was 2.2 ± 14.6 ml/min/1.73 m2. In the NOCTET trial, which comprised 282 Scandinavian heart and lung transplant recipients who were randomized to treatment with a CNI or low-dose CNI and everolimus 1-10 years after surgery, the measured glomerular filtration rate (GFR) declined 7.2 ml/min/1.73m2 during a mean follow up of 5.6 years (i.e. 1.3 ml/min/1.73m2 per year) independently of the time since transplantation and baseline GFR.

Proteinuria is an important determinant of ensuing renal failure. Approximately 25 % of patients listed for heart transplant have at least trace proteinuria. Of the investigators' maintenance heart transplant recipients, 18 % have manifest proteinuria defined as urine protein/creatinine ratio ≥ 30 mg/g. The median ratio is 49.5 mg/g (interquartile range 37-84), consistent with a daily loss of approximately 500 mg of protein in the urine.

Sodium-glucose cotransporter-2 inhibitors (SGLT2i) inhibit glucose reuptake in the proximal tubules of the nephrons. They thereby cause loss of glucose in the urine and induce osmotic diuresis. SGLT2i have now been studied in several large placebo-controlled cardiovascular outcomes trials in patients with type 2 diabetes. These trials were performed to satisfy regulatory requirements, specifically to exclude the excess risk of cardiovascular death, myocardial infarction, or stroke, and to test for efficacy. Despite a modest reduction in glycated haemoglobin (HbA1c), all the trials so far have shown that SGLT2i robustly reduces the risk of hospitalization for heart failure and prevents the progression of kidney disease.

In the EMPA-REG OUTCOME trial, treatment with the SGLT-2 inhibitor empagliflozin resulted in a reduction of cardiovascular mortality of 38%. In addition, empagliflozin significantly reduced admissions for heart failure and the incidence of end-stage kidney disease. Among patients allocated to empagliflozin, the mean change in estimated GFR (eGFR) from baseline to follow-up after 3 years was 4.7 ml per minute per 1.73 m2 better than in patients allocated to placebo. However, immediately after starting the drug, the patients on active treatment experienced an apparent reduction in the eGFR. The curves did not cross until after the first year of treatment, where after a between-group difference was manifest in favor of empagliflozin. The event curves diverged right up to the end of the trial, and there was an additional increase in the difference in the eGFR between the active drug arm and the placebo arm after stopping the treatment, suggesting that while empagliflozin is indeed renoprotective in patients with type 2 diabetes, there is an on-treatment suppression of eGFR analogue to the effect produced by angiotensin-converting enzyme inhibitors/angiotensin II receptor antagonists.

The DECLARE-TIMI 58 trial showed that the SGLT-2 inhibitor dapagliflozin reduced the rate of cardiovascular death or hospitalization for heart failure in a manner consistent with the findings observed in the EMPA-REG trial. Dapagliflozin was also associated with a large reduction in the rate of progression to end-stage renal failure. In consistence with the data on empagliflozin, 6 months after randomization, the mean decrease in the estimated GFR was larger in the dapagliflozin group than in the placebo group. However, the mean change equalized by 2 years, and at 3 and 4 years the mean decrease in eGFR was less with dapagliflozin than with placebo. The absolute difference in eGFR was smaller than that observed in the EMPA-REG OUTCOMES trial; however, the inclusion criteria in the DECLARE-TIMI 58 trial ensured that most of the participants had normal kidney function at the start of the treatment period. In the CREDENCE trial, canagliflozin had a similar effect on the glomerular filtration rate with the curves crossing at approximately one year. The effect on proteinuria, on the other hand, was substantial, occurred soon after the start of treatment, and was sustained for the entire study period. In the randomized, double-blind DELIGHT trial, dapagliflozin reduced the urine albumin-to-creatinine ratio in type 2 diabetics with 21.0 % (95 % confidence interval -34.1 to -5.2; p=0.01) after 24 weeks of treatment. The effect was almost immediate and was sustained from 4-24 weeks.

Several facts suggest that the cardioprotective and renoprotective effects of SGLT-2 inhibitors are to some extent independent of their glucose-lowering effect. First, the reductions in the levels of HbA1c in the EMPA-REG OUTCOMES and DECLARE TIMI 58 trials were modest compared with the pronounced effects on cardiovascular and renal outcomes. Second, the effect on renal outcomes seems to be independent of the effect on HbA1c. Third, the DAPA-HF trial in patients with and without diabetes recently demonstrated that the effect on cardiovascular outcomes was as large in non-diabetics as in patients with diabetes. Finally, in the DAPA-CKD trial, 4304 patients with a baseline eGFR between 25 and 75 ml/min/1.73m2 with or without diabetes were randomized to treatment with dapagliflozin 10 mg or placebo once daily. The primary endpoint was a sustained decline in eGFR ≥ 50 %, end-stage kidney disease, or renal or cardiovascular death. There was a substantial reduction in the hazard of reaching the primary endpoint in the dapagliflozin arm (hazard ratio 0.61, p < 0.001) irrespective of whether the patients had diabetes or not.

One of the major mechanisms of action of the SGLT-2 inhibitors is to decrease proximal tubular sodium and chloride reabsorption in the kidneys, leading to a reset of the tubuloglomerular feedback. This induces plasma volume contraction without activation of the sympathetic nerve system, decreases harmful glomerular hyper-filtration leading to better long-term renal preservation, and improves the diuretic and natriuretic responses to other diuretic agents. How this translates into a beneficial effect on the cardiovascular system is at present unclear. Heart transplant recipients have many common features with the heart failure population with metabolic disturbances, a propensity for coronary disease (allograft vasculopathy), and progressive nephropathy. Based on these premises, DAPARHT trial is designed to assess the hypothesis that treatment with dapagliflozin for one year ameliorates the decline in kidney function that often occurs in heart transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Heart transplant recipient ≥ 1 year after heart transplant.
2. Age ≥ 18 years

Exclusion Criteria:

1. Contraindications to study medication.
2. Estimated GFR < 25 ml/min/m2
3. Type I diabetes
4. Severe liver failure (Child-Pugh's score C)
5. Life expectancy reduced to < 2 years as judged by the investigator
6. Unresolved malignant disease
7. Failure to obtain written informed consent
8. SGL2 inhibitor treatment over the last month
9. Pregnancy
10. Breast-feeding
11. Woman of child-bearing potential who is not willing to use a highly effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
The chronic slope of the eGFR | From 2 weeks to end-of-treatment (12 months)
  The primary endpoint will be the slope of the eGFR from 2 weeks to end-of-treatment (12 months), calculated as the difference in eGFR from two weeks to 12 months after start of the intervention.

SECONDARY OUTCOMES:
Body weight | From 2 weeks to end-of-treatment (12 months)
  Change in body weight 2. The change in the albumin / creatinine ratio in the urine from baseline to end-of-treatment in patients with a baseline ratio > 30 mg/g at baseline 3. The change in the blood level of glycated haemoglobin (HbA1c) in patients with diabetes mellitus
Glycosylated hemoglobin (HbA1c) | From 2 weeks to end-of-treatment (12 months)
  Change in the blood level of HbA1c in patient with diabetes mellitus
Proteinuria | From 2 weeks to end-of-treatment (12 months)
  Change in the albumin / creatinine ratio in the urine in patients with a baseline ratio > 30 mg/g

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Manintveld, MD, PhD, Principal Investigator — Erasmus Medical Center; Oscar Braun, MD, PhD, Principal Investigator — Skane University Hospital; Ida H Löfman, MD, PhD, Principal Investigator — Karolinska University Hospital; Kevin Damman, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (6):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam
- Oslo University Hospital, Rikshospitalet, Oslo, Oslo County, Norway
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmen S, Manintveld O, Damman K, Braun O, Lofman IH, Szymanski M, Ravnestad H, Gude E, Bjorkelund E, Andreassen AK, Gullestad L, Broch K. DAPAgliflozin for renal protection in heart transplant recipients. Rationale and design of the randomized controlled DAPARHT trial. Am Heart J. 2026 Jan;291:128-135. doi: 10.1016/j.ahj.2025.08.010. Epub 2025 Aug 19. PMID 40840822
- [Derived] Garcia-Cosio Carmena MD, Farrero M, Blasco Peiro MT, Crespo M, Delgado Jimenez J, Diaz Molina B, Fernandez Rivera C, Garrido Bravo IP, Lopez Jimenez V, Melilli E, Mirabet Perez S, Perez Tamajon ML, Rangel Sousa D, Rodrigo E, Cruzado JM, Hernandez Marrero D; Spanish Society of Transplantation, the Spanish Society of Nephrology, and the Spanish Society of Cardiology (SET-SEC-SEN). Management of Kidney Disease in Heart Transplant Patients: A National Delphi Survey-based Consensus Expert Paper. Transplantation. 2025 Sep 1;109(9):e431-e445. doi: 10.1097/TP.0000000000005302. Epub 2025 Feb 7. PMID 39928546